CLINICAL TRIAL: NCT02042352
Title: PNA FISH, PCR and Gram Staining for Detection of Bacterial Vaginosis - a Comparative Clinical Study in a Danish IVF Setting
Status: Completed | Type: Observational
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Other Study IDs: RSkive
Record Dates: First submitted 2014-01-16; First posted 2014-01-22 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal flora swabs

GROUPS / COHORTS (1):
- pH test: VpH test gloves
  Interventions: Other: pH glove

INTERVENTIONS:
Other: pH glove

SUMMARY:
The primary aim of the present study is to investigate the vaginal microbiota of infertile women with two novel molecular based diagnostic tests for Bacterial Vaginosis, a PNA FISH and a PCR method supported with conventional Gram staining.

We hypothesize that the molecular based tests will prove more efficient than conventional Gram staining and that they have a place in future IVF diagnostics.

DETAILED DESCRIPTION:
Our first aim is to investigate the prevalence of altered vaginal microbiotas among women seeking fertility treatment in Denmark. Secondly we want to establish whether there are correlations between altered vaginal microbiotas and self-measurements of both the vaginal pH performed with the Saling pH glove™ and a self-collected swab with Copan Eswab™ because these would be useful for an easy-access longitudinal screening option. Finally, the third aim was to explore how the species composition of vaginal microbiotas measured by a multiplex qPCR assay was reflected in Nugent scores.

A possible 4th aim is to identify patterns in the relative abundances of different species with 16sRNA primers among fertile women compared with infertile women because these differences could be indicative of a vaginal microbiota associated with bad fertility outcome.

ELIGIBILITY:
Inclusion Criteria:

* Seeking IVF treatment

Exclusion Criteria:

* Bleeding and sexual intercourse within 24h

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IVF patients
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cost-benefit analysis of the molecular tests to conventional Gram staining | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic Skive, Skive, Denmark

REFERENCES:
- [Derived] Jakobsen RR, Haahr T, Humaidan P, Jensen JS, Kot WP, Castro-Mejia JL, Deng L, Leser TD, Nielsen DS. Characterization of the Vaginal DNA Virome in Health and Dysbiosis. Viruses. 2020 Oct 9;12(10):1143. doi: 10.3390/v12101143. PMID 33050261
- [Derived] Haahr T, Humaidan P, Elbaek HO, Alsbjerg B, Laursen RJ, Rygaard K, Johannesen TB, Andersen PS, Ng KL, Jensen JS. Vaginal Microbiota and In Vitro Fertilization Outcomes: Development of a Simple Diagnostic Tool to Predict Patients at Risk of a Poor Reproductive Outcome. J Infect Dis. 2019 May 5;219(11):1809-1817. doi: 10.1093/infdis/jiy744. PMID 30597027
- [Derived] Haahr T, Jensen JS, Thomsen L, Duus L, Rygaard K, Humaidan P. Abnormal vaginal microbiota may be associated with poor reproductive outcomes: a prospective study in IVF patients. Hum Reprod. 2016 Apr;31(4):795-803. doi: 10.1093/humrep/dew026. Epub 2016 Feb 23. PMID 26911864